CLINICAL TRIAL: NCT00722631
Title: Detection of Plaque Inflammation and Visualization of Anti-Inflammatory Effects of Pioglitazone on Plaque Inflammation in Subjects With Impaired Glucose Tolerance and Type 2 Diabetes Mellitus by FDG-PET/CT
Brief Title: Anti-Inflammatory Effects of Pioglitazone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Nobuhiro Tahara, M.D., PhD, Kurume University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIO 2007
Record Dates: First submitted 2008-07-22; First posted 2008-07-25 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Impaired Glucose Tolerance; Type 2 Diabetes Mellitus; Atherosclerosis
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): up to 30 mg pioglitazone, tablet, orally, once daily
  Interventions: Drug: Pioglitazone
- 2 (Active Comparator): up to 4 mg/day glimepiride, tablet, orally, once daily
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Pioglitazone — Subjects who meet eligibility criteria will be titrated up to a maximum of 30 mg/day pioglitazone.
  Other Names: CAS number: 111025-46-8, ATC code: A10BG03
  Arms: 1
Drug: Glimepiride — Subjects who meet eligibility criteria will be titrated up to a maximum of 4 mg/day glimepiride.
  Other Names: CAS number: 93479-97-1, ATC code: A10BB12
  Arms: 2

SUMMARY:
There is increasing evidence that inflammation plays a role in progression and destabilization of atherosclerotic plaque. FDG-PET can visualize activated metabolic activity of inflammatory cells. It is possible that FDG-PET can detect atherosclerotic plaque inflammation and that FDG-PET can monitor the effect of pioglitazone on plaque inflammation.

DETAILED DESCRIPTION:
Atherosclerotic patients with impaired glucose tolerance and type 2 diabetes will undergo the FDG-PET/CT imaging at baseline and again following 4 months after treatment. Patients who meet eligibility criteria will be titrated up to a maximum of 30 mg/day pioglitazone or 4 mg/day glimepiride. Physical examinations will be done at baseline, 4 months, and 12 months. During study, subjects will have body weight, and vital signs (HR, BP, etc) assessed as well as waist circumference. Laboratory assessments will be done at each baseline, 4 month.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 35 and 85 years
* Subjects with impaired glucose tolerance and type 2 diabetes, who had atherosclerosis detected by carotid ultrasound and/or CT
* Subjects who had vascular FDG uptake by FDG-PET

Exclusion Criteria:

* Subjects with insulin treatment
* Subjects with uncontrolled diabetes, hypertension, symptomatic coronary artery disease, symptomatic cerebrovascular disease
* Subjects taking more than three antidiabetic medications
* Subjects taking anti-platelet, statins, antidiabetic agents, thiazolidinediones (TZDs) within 8 weeks prior to randomization
* Subjects with cardiac failure (New York Heart Association Class > III) or left ventricular dysfunction (LVEF < 40%)
* Subjects with systemic disorders such as active inflammatory, liver, renal, hematopoietic, and malignant disease

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on the nominal change in FDG uptake of atherosclerotic plaque from baseline after 4 months of treatment as measured by FDG-PET/CT imaging. | Baseline and 4 months after treatment

SECONDARY OUTCOMES:
Change from baseline in plasma glucose/insulin homeostatic parameters and circulating markers of atherosclerosis | Baseline and 4 months and 5 years after treatment
Change from baseline in visceral fat | Baseline and 4 months and 5 years after treatment
All cardiovascular events and all cause death for 5 years | Baseline and 4 months and 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhiro Tahara, MD, PhD, Principal Investigator — Kurume University
Locations (1):
- Kurume University Hospital, Kurume, Japan

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751
- [Derived] Tahara N, Nitta Y, Bekki M, Tahara A, Maeda-Ogata S, Sugiyama Y, Honda A, Igata S, Nakamura T, Sun J, Kurata S, Fujimoto K, Abe T, Matsui T, Yamagishi SI, Fukumoto Y. Two-hour postload plasma glucose and pigment epithelium-derived factor levels are markers of coronary artery inflammation in type 2 diabetic patients. J Nucl Cardiol. 2020 Aug;27(4):1352-1364. doi: 10.1007/s12350-019-01842-5. Epub 2019 Aug 12. PMID 31407236
- [Derived] Nitta Y, Tahara N, Tahara A, Honda A, Kodama N, Mizoguchi M, Kaida H, Ishibashi M, Hayabuchi N, Ikeda H, Yamagishi S, Imaizumi T. Pioglitazone decreases coronary artery inflammation in impaired glucose tolerance and diabetes mellitus: evaluation by FDG-PET/CT imaging. JACC Cardiovasc Imaging. 2013 Nov;6(11):1172-82. doi: 10.1016/j.jcmg.2013.09.004. PMID 24229770
- [Derived] Kodama N, Tahara N, Tahara A, Honda A, Nitta Y, Mizoguchi M, Kaida H, Ishibashi M, Abe T, Ikeda H, Narula J, Fukumoto Y, Yamagishi S, Imaizumi T. Effects of pioglitazone on visceral fat metabolic activity in impaired glucose tolerance or type 2 diabetes mellitus. J Clin Endocrinol Metab. 2013 Nov;98(11):4438-45. doi: 10.1210/jc.2013-2920. Epub 2013 Sep 12. PMID 24030946
- [Derived] Mizoguchi M, Tahara N, Tahara A, Nitta Y, Kodama N, Oba T, Mawatari K, Yasukawa H, Kaida H, Ishibashi M, Hayabuchi N, Harada H, Ikeda H, Yamagishi S, Imaizumi T. Pioglitazone attenuates atherosclerotic plaque inflammation in patients with impaired glucose tolerance or diabetes a prospective, randomized, comparator-controlled study using serial FDG PET/CT imaging study of carotid artery and ascending aorta. JACC Cardiovasc Imaging. 2011 Oct;4(10):1110-8. doi: 10.1016/j.jcmg.2011.08.007. PMID 21999871